CLINICAL TRIAL: NCT05931861
Title: Performance and Safety Assessment of T2769 in Contact Lens Wearers With Dry Eye Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT2769-003
Record Dates: First submitted 2023-06-23; First posted 2023-07-05 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T2769 (Experimental): One drop in each eye, from 3 to 6 times daily, at any time but only when patients are wearing their contact lenses.
  Interventions: Device: T2769

INTERVENTIONS:
Device: T2769 — T2769: sodium hyaluronate 0.15%, Trehalose 3%, Naaga 2.45% in a 12.5 mL ABAK® multi-dose bottle.

SUMMARY:
This is a confirmatory clinical investigation. The objective is to collect new additional clinical data demonstrating the safety and performance of the device in the contact-lens wearing population with dry eyes. The hypotheses are that T2769 improves dry eye symptomatology (e.g. decrease in CLDEQ-8 score, in OSDI score, ocular discomfort assessed by VAS) and signs (e.g. increase in Schirmer and TBUT, decrease in Oxford score) at D36, in comparison to baseline.

The primary objective of this investigation is to assess the performance of T2769 in contact lens wearers with dry eye symptoms in terms of change from baseline (Day 1) to Day 36 (Final visit) in Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) total score.

ELIGIBILITY:
Main Inclusion Criteria:

* Informed consent signed and dated
* Patient aged ≥ 18 years old
* Well fitted contact lenses (CL) according to the investigator judgement
* Daily wearer of any type of CL for a minimum of 5 days/week for 6 hours/day over at least the last month and is willing to continue to do so during the study
* Patient with an Ocular Surface Disease Index (OSDI) score ≥ 18
* CLDEQ-8 score ≥ 12

Main Exclusion Criteria:

* Far Best-Corrected Visual Acuity (BCVA) ≥+0.7 LogMar (e.g., ≤0.2 in decimal value or ≤20/100 Snellen equivalent or ≤50 ETDRS letters).
* Severe blepharitis
* Severe Meibomian gland dysfunction
* Palpebral or nasolacrimal disorders
* Dry eye associated with at least one of the following diseases/symptoms: ocular rosacea, Pterygium, Eyelid malposition, Corneal dystrophy, Ocular neoplasia, Filamentous keratitis, Corneal neovascularisation, Orbital radiotherapy, Cataract, Retinal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Grupcheva, Professor, Principal Investigator — Individual Practice for Specialized Ophthalmology Care
Locations (6):
- Bulgaria (6):
  - Medical Center "Oxycom", Burgas
  - "Asmp Ob - Ip Glm" Eood, Smolyan
  - Medical Center For Eye Health "Focus", Sofia
  - Specialized Ophthalmological Hospital For Active Treatment "Pentagram", Sofia
  - Medical Center "Vereya", Stara Zagora
  - Ambulatory For Group Practice For Specialized Medical Care For Eye Diseases - Dr. Grupchevi, Varna

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2769
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | T2769
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Total Score.
Description: The primary endpoint is the change from baseline (Day 1) to Day 36 in the Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) total score.
  CLDEQ-8 consists of 8 questions designed to measure dry eye symptoms specifically related to the use of contact lenses. The total score is obtained by adding the scores obtained for each answer. The final score is ranging from 1 to 37.
  37 is the worst score.
Time Frame: CLDEQ- score is assessed at Day 1 and Day 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T2769
Number analyzed (Participants) | 34
score on a scale | -12.6 (5.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent signature (Day 1) to Final visit (Day 36).
Arm/Group | T2769
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data resulting from this clinical investigation will be the proprietary information of Sponsor. An investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with Laboratoires THÉA in advance.

DOCUMENTS (2):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT05931861/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05931861/SAP_001.pdf